CLINICAL TRIAL: NCT00119522
Title: Epidemiology and Cost of Falls in Veterans With Spinal Cord Injury
Brief Title: Epidemiology and Cost of Falls in Veterans With a Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 03-003
Record Dates: First submitted 2005-07-01; First posted 2005-07-13 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-07

CONDITIONS: Spinal Cord Injury
Keywords: wheelchairs; falls; spinal cord injury; accidental falls; safety
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: cohort is of individuals with a spinal cord injury who use a wheelchair as their primary means of mobility

SUMMARY:
Brief Summary Detailed Description Background: A multitude of risk factors for falling has been reported for the elderly, however many of these risk factors are not applicable to persons with a spinal cord injury, who use a wheelchair for mobility. The objectives of this study are to: (1) describe the incidence and prevalence of tips, falls, and fall-related injuries in SCI; (2) describe the epidemiology of the fall event (person, time, place, and activity); (3) describe any injuries associated with a fall, including the mechanism and nature of the injury, severity of injury, as well as treatment required; (4) determine the risk factors related to falls and fall-related injuries in SCI, and develop a model for predicting falls and fall-related injuries in SCI; (5) determine healthcare utilization as well as direct and indirect costs associated with fall-related injuries in SCI; and (6) describe patient-perceived short- and long-term consequences of falls in SCI. The data collection for this study was completed on March 31, 2007, and data analysis is in final phase.

Objectives: The objectives of the study are to describe: (1) the incidence and prevalence of wheelchair tips, falls, and fall-related injuries; (2) epidemiology of event; (3) injuries associated with event, including mechanism, nature, severity of injury and treatment required; (4) determine risk factors and develop a model for predicting tips and falls; (5) determine healthcare utilization and direct and indirect costs; and (6) describe perceived short- and long-term consequences of falls in SCI.

Methods: This is a prospective cohort study. Data was collected through patient surveys, medical records, and VA databases. Baseline information includes risk factors (e.g., user characteristics, wheelchair features, wheelchair activities, etc.) and physical environmental data. Monthly follow-up calls tracked tips, falls, and injuries.

Status: Recruitment ended on April 1, 2006 with a total of 702 subjects, and data collection was completed on March 31, 2007. The Data Safety Monitoring Board for this study conducted its final meeting on September 17, 2007. Data has been analyzed and 17 manuscripts are currently in development.

Impact: While much is known about falls in elderly, there is a lack of understanding of the epidemiology of wheelchair-related falls. Our project is expected to identify previously unaccounted for factors that predispose persons with SCI to falls and fall-related injuries. This study will result in the creation of a model for predicting falls and fall-related injuries in SCI. The predictive model will be used to develop intervention strategies targeting modifiable risk factors. Eventually, we will test this predictive model with other vulnerable veteran populations. Findings from this study wil be used to develop an instrument to identify fall risk in persons with SCI.

DETAILED DESCRIPTION:
Of the 702 patients enrolled, 659 subjects provided data for follow up analysis. The primarily male (96%) population was 55 + 13 years old, and had their SCI for an average of 21 + 13 years. 47% of the injury levels were cervical and 46% thoracic. The majority of subjects used manual wheelchairs (62%) an average of 10.9 + 4.3 hours a day. 553 fall events were reported by 204 individuals. 95 (14%) subjects were injured as a result of the fall. Regression models showed that fall occurrence was predicted by increased pain in past two months, increased alcohol use, higher FIM sub-motor scores, having a previous fall, shorter wheelchair length, fewer years of SCI, and not having one's first wheelchair. Injurious falls were predicted by increased pain in past two months, higher FIM sub-motor scores, having a previous fall, non-flat home entrance and a diagnosis of arthritis. In both models, 83% of the variance was explained by the predictors. Additional analysis is planned for completion of manuscripts. In addition, funding was received to develop a risk assessment tool for falls from wheelchairs in SCI.

Final analyses are being conducted and 17 manuscripts are currently in development.

ELIGIBILITY:
Inclusion Criteria:

Must be a veteran with a spinal cord injury and use a wheelchair as primary means of mobility.

Exclusion Criteria:

Spinal cord injury less than 2 years. Use of mobility device other than wheelchair as primary means of mobility. Incomplete injury that does not warrant use of a wheelchair. Ventilator dependent. On bedrest for more than 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: spinal cord injury population
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2004-04; Primary Completion 2006-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
tips and falls from wheelchairs | one year

CONTACTS AND LOCATIONS:
Overall Officials: Audrey L. Nelson, RN PhD FAAN, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (3):
- United States (3):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Charlie Norwood VA Medical Center, Augusta, GA, Augusta, Georgia
  - VA Boston Healthcare System Brockton Campus, Brockton, MA, Brockton, Massachusetts

REFERENCES:
- [Result] Gavin-Dreschnack D, Nelson A, Fitzgerald S, Harrow J, Sanchez-Anguiano A, Ahmed S, Powell-Cope G. Wheelchair-related falls: current evidence and directions for improved quality care. J Nurs Care Qual. 2005 Apr-Jun;20(2):119-27. doi: 10.1097/00001786-200504000-00006. PMID 15839290
- [Result] Gavin-Dreschnack D. Effects of wheelchair posture on patient safety. Rehabil Nurs. 2004 Nov-Dec;29(6):221-6. PMID 15598002
- [Result] Nelson AL, Groer S, Palacios P, Mitchell D, Sabharwal S, Kirby RL, Gavin-Dreschnack D, Powell-Cope G. Wheelchair-related falls in veterans with spinal cord injury residing in the community: a prospective cohort study. Arch Phys Med Rehabil. 2010 Aug;91(8):1166-73. doi: 10.1016/j.apmr.2010.05.008. PMID 20684896